CLINICAL TRIAL: NCT02927964
Title: Intratumoral Injection of SD-101, an Immunostimulatory CpG, in Combination With Ibrutinib and Local Radiation in Relapsed or Refractory Low-Grade Follicular Lymphoma
Brief Title: TLR9 Agonist SD-101, Ibrutinib, and Radiation Therapy in Treating Patients With Relapsed or Refractory Grade 1-3A Follicular Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Lowsky (Other)
Collaborators: Janssen, LP (Industry); National Cancer Institute (NCI) (NIH); The Leukemia and Lymphoma Society (Other); Rising Tide Foundation (Other)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-36750; NCI-2016-01065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-36750 (Other: Stanford IRB); LYMNHL0135 (Other: OnCore); R35CA197353 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2023-09

CONDITIONS: Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Recurrent Follicular Lymphoma; Refractory Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — ibrutinib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1b -SD-101 3mg (Experimental): Patients undergo radiation therapy on days 1 and 2. Within 12 hours of the completion of radiation therapy, patients receive TLR9 agonist SD-101 IT on day 2 and on days 9, 16, 23, 30 and 37. Patients also receive ibrutinib PO daily beginning on day 9 for 96 weeks or in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Ibrutinib; Radiation: Radiation Therapy; Drug: TLR9 Agonist SD-101

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; PCI-32765
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: TLR9 Agonist SD-101 — Given IT
  Other Names: ISS-ODN SD-101; SD-101

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of toll-like receptor 9 (TLR9) agonist SD-101 when given together with ibrutinib and radiation therapy and to see how well they work in treating patients with Low Grade Follicular Lymphoma, Marginal Zone Lymphoma, or Mantle Cell Lymphoma that has come back after a period of improvement or no longer responds to treatment. Immunostimulants such as TLR9 agonist SD-101 may increase the ability of the immune system to fight infection and disease. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving TLR9 agonist SD-101 with ibrutinib and radiation therapy may induce an immune response and prolong anti-tumor response.

DETAILED DESCRIPTION:
Primary Objective:

Phase 1b: - To determine the recommended phase 2 dose (RP2D) of intratumoral SD 101 in combination with ibrutinib and radiation in subjects with relapsed or refractory B cell lymphoma . - To determine the safety and tolerability of SD 101 in combination with ibrutinib and radiation in subjects with relapsed or refractory B cell lymphoma

Phase 2: -To evaluate the efficacy of intratumoral SD 101 in combination with ibrutinib and radiation in subjects with relapsed or refractory B cell lymphoma by assessing overall response rate

Secondary Objective:

Phase 2: - To evaluate progression free survival after treatment with intratumoral SD 101 in combination with ibrutinib and radiation in subjects with relapsed or refractory B cell lymphoma

- To evaluate the induction of tumor-specific immune responses by treatment with intratumoral SD-101 in combination with ibrutinib and radiation in patients with relapsed or refractory B cell lymphoma

ELIGIBILITY:
Inclusion Criteria

* Biopsy confirmed Grade 1 or 2, or 3A follicular lymphoma; mantle cell lymphoma; or marginal zone lymphoma. Subjects must have relapsed from or are refractory to prior therapy.
* Subjects must have at least one site of disease that is accessible for intratumoral injection of SD 101 (diameter ≥ 10mm), percutaneously.
* Subjects must have at least one site of measurable disease (see Section 10.2.2 for definition of measurable disease) other than the injection site which is not included in the radiation field.
* ECOG Performance Status of 0 or 1
* Subjects must be 18 years of age or older.
* Required values for initial laboratory tests:

  1. Absolute neutrophil count (ANC) ≥ 1000/mm3 independent of growth factor support
  2. Platelets: ≥ 100,000/mm3 or ≥ 50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
  3. Hemoglobin: ≥ 8 g/dL (may be transfused)
  4. Creatinine: Creatinine clearance > 25 mL/min
  5. AST/ALT: ≤ 3 x ULN
  6. Bilirubin: ≤ 1.5 x ULN (except for subjects with Gilbert's Syndrome or of non hepatic origin)
* Must be at least 4 weeks since treatment with standard or investigational chemotherapy, biochemotherapy, surgery, radiation, cytokine therapy, and 8 weeks since any monoclonal antibodies or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment.
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Life expectancy greater than 4 months.
* Able to comply with the treatment schedule.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Autoimmune disease requiring treatment within the last 5 years including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjӧgren's syndrome, autoimmune thrombocytopenia, uveitis, or other if clinically significant
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists.
* Requires chronic treatment with strong CYP3A inhibitors.
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment.
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection.
* Known CNS lymphoma.
* Subjects with a history of prior malignancy with the exception of non melanoma skin cancer, carcinoma in situ of the cervix, in situ carcinoma of the bladder, stage 1 prostate cancer that does not require treatment, or other malignancy that has undergone potentially curative therapy with no evidence of disease for the last > 2 years and that is deemed by the investigator to be a low risk for recurrence.
* History of allergic reactions attributed to compounds of similar composition to SD 101 or ibrutinib
* Treatment with an immunosuppressive regimen of corticosteroids or other immunosuppressive medication (eg, methotrexate, rapamycin) within 30 days of study treatment. Note: subjects may take up to 5 mg of prednisone or equivalent daily. Topical and inhaled corticosteroids in standard doses are allowed.
* Significant cardiovascular disease (ie, NYHA class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Pregnant or breast feeding.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University; Michael Khodadoust, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Derived] Shree T, Haebe S, Czerwinski DK, Eckhert E, Day G, Sathe A, Grimes S, Frank MJ, Maeda LS, Alizadeh AA, Advani R, Hoppe RT, Long SR, Martin B, Ozawa MG, Khodadoust MS, Ji HP, Levy R. A clinical trial of therapeutic vaccination in lymphoma with serial tumor sampling and single-cell analysis. Blood Adv. 2024 Jan 9;8(1):130-142. doi: 10.1182/bloodadvances.2023011589. PMID 37939259
- [Derived] Mooney KL, Czerwinski DK, Shree T, Frank MJ, Haebe S, Martin BA, Testa S, Levy R, Long SR. Serial FNA allows direct sampling of malignant and infiltrating immune cells in patients with B-cell lymphoma receiving immunotherapy. Cancer Cytopathol. 2022 Mar;130(3):231-237. doi: 10.1002/cncy.22531. Epub 2021 Nov 15. PMID 34780125

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I -SD-101 3mg; Phase II -SD-101 3mg: Patients underwent radiation therapy on days 1 and 2. Within 12 hours of the completion of radiation therapy, patients received TLR9 agonist SD-101 IT on day 2 and on days 9, 16, 23, 30 and 37. Patients also received ibrutinib PO daily beginning on day 9 for 96 weeks or in the absence of disease progression or unexpected toxicity.
Period: Overall Study
Arm/Group | Phase I -SD-101 3mg | Phase II -SD-101 3mg
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib); Phase II -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib): Patients underwent radiation therapy on days 1 and 2. Within 12 hours of the completion of radiation therapy, patients received TLR9 agonist SD-101 IT on day 2 and on days 9, 16, 23, 30 and 37. Patients also received ibrutinib PO daily beginning on day 9 for 96 weeks or in the absence of disease progression or unexpected toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1b -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) | Phase II -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicity Assessed Using Common Terminology Criteria for Adverse Events Version 4.0 (Phase Ib)
Description: Dose-limiting toxicity was continuously throughout the trial. Adverse event information was collected at each visit. Safety labs were collected on week 2, 4, 6, 12 and every 12 weeks thereafter until the final study visit.
Time Frame: Up to 24 months
Population: Participants who received treatment are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) | Phase II -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib)
Number analyzed (Participants) | 6 | 0
Participants | 1 | 0

2. Primary Outcome: Tumor Response Rates (Phase II)
Description: Tumor response rate of intratumoral SD 101 in combination with ibrutinib and radiation in subjects will be assessed. Tumor response rates (complete response, partial response) will be calculated based on the Lugano classification for low-grade B-cell lymphomas.
Time Frame: Up to 24 months
Population: Participants who received treatment are included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib); Phase II -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib): Patients underwent radiation therapy on days 1 and 2. Within 12 hours of the completion of radiation therapy, patients received TLR9 agonist SD-101 IT on day 2 and on days 9, 16, 23, 30 and 37. Patients also received ibrutinib PO daily beginning on day 9 for 96 weeks or in the absence of disease progression or unexpected toxicity.
Arm/Group | Phase 1b -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) | Phase II -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib)
Number analyzed (Participants) | 11 | 9
Participants
  Complete Response | 0 | 1
  Partial Response | 4 | 5

3. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression free Survival is defined as the time elapsed between treatment initiation (Day 1) and tumor progression or death from any cause. Progression will be defined using the Lugano Classification. This outcome will be measured on any individual who has received at least one intratumoral injection of SD 101 at the recommended phase 2 dose level.
Time Frame: Up to 24 months
Population: Participants who received treatment are included in the analysis
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase 1b -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) | Phase II -SD-101 3mg:Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib)
Number analyzed (Participants) | 11 | 9
Months | 11 [7.0 to 21.9] | 11 [7.0 to 21.9]

ADVERSE EVENTS:
Time Frame: up to 24 months
Groups:
- Phase 1b/phase2 -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib): Patients underwent radiation therapy on days 1 and 2. Within 12 hours of the completion of radiation therapy, patients received TLR9 agonist SD-101 IT on day 2 and on days 9, 16, 23, 30 and 37. Patients also received ibrutinib PO daily beginning on day 9 for 96 weeks or in the absence of disease progression or unexpected toxicity.
Arm/Group | Phase 1b/phase2 -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b/phase2 -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) (N=20)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
maculopapular rash (Skin and subcutaneous tissue disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Infection other (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b/phase2 -SD-101 3mg: Treatment (Radiation Therapy, TLR9 Agonist SD-101, Ibrutinib) (N=20)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Palpitations (Cardiac disorders) | 6 (7)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 3 (3)
Eye Pain (Eye disorders) | 3 (3)
Dry Eyes (Eye disorders) | 1 (1)
Eye Infection (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 16 (34)
Nausea (Gastrointestinal disorders) | 11 (28)
Abdominal Pain (Gastrointestinal disorders) | 9 (14)
Oral mucositis (Gastrointestinal disorders) | 7 (14)
Dyspepsia (Gastrointestinal disorders) | 8 (10)
Sore Throat (Gastrointestinal disorders) | 4 (13)
Dry mouth (Gastrointestinal disorders) | 4 (5)
Bloating (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
Dysgeusia (Gastrointestinal disorders) | 3 (3)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Bleeding gum (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dark stool (Gastrointestinal disorders) | 1 (1)
Early satiety (Gastrointestinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Swollen lip (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 19 (49)
Injection site reaction (General disorders) | 15 (40)
Chills (General disorders) | 15 (37)
Fever (General disorders) | 11 (22)
Edema limbs (General disorders) | 2 (5)
Malaise (General disorders) | 3 (3)
Chest pain (General disorders) | 4 (8)
Ear pain (General disorders) | 1 (1)
General pain (General disorders) | 2 (2)
Naval pain (General disorders) | 1 (1)
Neck pain (General disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 6 (8)
Skin infection (Infections and infestations) | 3 (6)
Bronchial infection (Infections and infestations) | 3 (3)
Bursitis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Skin wound (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 12 (15)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 1 (2)
Shoulder injury (Injury, poisoning and procedural complications) | 1 (1)
Arm injury (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (18)
White blood cell count decreased (Investigations) | 9 (12)
Neutrophil count decreased (Investigations) | 6 (11)
Creatinine increased (Investigations) | 3 (4)
Increased LDH (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase decreased (Investigations) | 1 (1)
Monocyte increased (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Chloride increased (Investigations) | 1 (1)
Low Chloride (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
High ketones (Investigations) | 1 (1)
Low magnesium (Investigations) | 1 (1)
Low Phosphorus (Investigations) | 1 (1)
Low Ferritin (Investigations) | 1 (1)
Low serum globulin concentration (Investigations) | 1 (1)
Low transferrin saturation (Investigations) | 1 (1)
Low Albumin (Investigations) | 1 (1)
High PTT (Investigations) | 1 (1)
Platelet count decreased (Metabolism and nutrition disorders) | 11 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (7)
Loss of appetite (anorexia) (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (20)
Back and shoulder pain (Musculoskeletal and connective tissue disorders) | 7 (17)
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 5 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 15 (58)
Dizziness (Nervous system disorders) | 4 (7)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3)
Lightheadedness (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Confusion (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Decreased libido (Psychiatric disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 11 (29)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (7)
Itchiness (Skin and subcutaneous tissue disorders) | 4 (6)
Night Sweats (Skin and subcutaneous tissue disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Dry brittle finger nails (Skin and subcutaneous tissue disorders) | 3 (3)
Blisters (Skin and subcutaneous tissue disorders) | 3 (3)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Bleeding (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (7)
Flushing (Vascular disorders) | 1 (1)
Cold hands and feet (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT02927964/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02927964/ICF_000.pdf